CLINICAL TRIAL: NCT02831257
Title: A Single Arm Phase 2 Study of the Dual mTORC1/mTORC2 Inhibitor AZD2014 Provided on an Intermittent Schedule for Neurofibromatosis 2 Patients With Progressive or Symptomatic Meningiomas
Brief Title: AZD2014 In NF2 Patients With Progressive or Symptomatic Meningiomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: AstraZeneca (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Scott R. Plotkin, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-590
Record Dates: First submitted 2016-07-07; First posted 2016-07-13 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Neurofibromatosis 2; Meningioma
Keywords: Neurofibromatosis 2
MeSH Terms: conditions — Neurofibromatosis 2; Meningioma | interventions — vistusertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD2014 (Experimental): 18 patients will be enrolled in this study in a single stage.
  * AZD2014 orally, 2 times a day on 2 consecutive day out of every 7 days.
  * One cycle will consist of 28 days (1 cycle = 28 days).
  Interventions: Drug: AZD2014

INTERVENTIONS:
Drug: AZD2014

SUMMARY:
The goal of this clinical research study is to learn if the study drug AZD2014 can shrink growing or symptomatic meningiomas.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The goal of this clinical research study is to learn if the study drug AZD2014 can shrink growing or symptomatic meningiomas. Based on laboratory research, the cellular pathways which are blocked by AZD2014 are important for the growth and survival of meningiomas. Further treatment of meningioma cells in the laboratory setting has resulted in decreased survival of tumor cells. As such, the purpose of this research is to see whether treating your meningioma with AZD2014 will result in tumor shrinkage. The safety of AZD2014 will also be studied. Your physical state, your symptoms, changes in the size of the tumor, and laboratory findings obtained while on-study will help the research team decide if AZD2014 is safe and effective in patients with your condition.

AZD2014 is being studied in patients with various cancers as a single agent (a drug that is used alone to treat the cancer) or in combination with a number of anticancer therapies. Previous studies have also allowed investigators to determine the best dose and frequency of AZD2014 to achieve anti-tumor effects while reducing the likelihood of side effects.

The FDA (the U.S. Food and Drug Administration) has not approved AZD2014 as a treatment for any disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of neurofibromatosis 2 by fulfilling National Institute of Health (NIH) criteria or Manchester criteria, or by detection of a causative mutation in the NF2 gene.
* Participants must have progressive or symptomatic meningioma. NOTE 1: Histologic confirmation of meningioma is not required in the setting of compatible radiographic appearance, NOTE2: progression is defined as an increase in target meningioma volume ≥ 20% OR ≥ 3 mm during the past 2 years.

  -- Subjects must have a target meningioma that is not amenable to surgery due to patient preference or high risk for surgical complications
* Participants must be willing and able to undergo regular MRI scans of the brain
* Patients must have measurable disease, defined as at least one meningioma ≥ 1.0 ml that can be accurately measured by contrast-enhanced cranial MRI scan, performed within 28 days of study registration.
* Prior surgical resection and radiation therapy for the progressive meningioma are not required for study enrollment.
* Patients must have received less than 3 prior chemotherapy regimens for progressive meningioma.
* Patients receiving dexamethasone must be able to be treated with alternative corticosteroids such as prednisone, prednisolone, or methylprednisolone in the opinion of the treating physician.
* Patients must have available an archival paraffin tumor block sufficient to generate at least 20 unstained slides; or, if a paraffin tumor block is unavailable, at least 20 unstained slides.
* Age ≥ 18 years at the time of study enrollment.
* ECOG performance status ≤2 (Karnofsky ≥60%) with no deterioration over the previous 2 weeks
* Life expectancy of greater than 3 months
* Within 14 days of study registration, participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * hemoglobin ≥90 g/L
  * platelets ≥100,000/mcL
  * total bilirubin ≤1.5 x institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * Serum creatinine ≤1.5 x institutional upper limit of normal concurrent with creatinine clearance ≥50 mL/min (measured or calculated by Cockcroft and Gault equation), confirmation of creatinine clearance is only required when creatinine is >1.5xULN
  * Urine protein ≤1+ on urine dipstick (if 2+ seen on first test, re-test at least 24 hours later)
  * PT/INR/PTT (aPTT) <1.5x institutional upper limit of normal
* The effects of AZD2014 on the developing human fetus are unknown. For this reason and because mTOR kinase inhibiting agents are known to be teratogenic, female patients must be willing to use 2 forms of highly effective contraception (per institution standards) from the time of screening until 4 weeks after discontinuing study, must not be breast feeding and must have a negative pregnancy test prior to start of dosing if of child bearing potential or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening: (1) post-menopausal women, defined as either women aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments, or, (2) women under 50 years old who have been amenorrhoeic for at least 12 months following the cessation of exogenous hormonal treatments, and have serum follicle-stimulating hormone (FSH) and luteinizing hormone (LH) levels in the postmenopausal range for the institution. Alternatively, women must have documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
* Male patients should either be surgically sterile or willing to use an effective barrier method of contraception during the study and for 16 weeks following the last dose of study treatment if sexually active with a female of childbearing potential. If not done previously, storage of sperm prior to receiving AZD2014 will be advised to male patients with a desire to have children.
* Ability to understand and the willingness to sign a written informed consent document prior to any study specific procedures, sampling, and analyses.
* Ability to swallow and retain oral medication

Exclusion Criteria:

* Prior chemotherapy, biological therapy, radiation therapy, androgens, thalidomide, immunotherapy, other anticancer agents within 21 days of starting study treatment (not including palliative radiotherapy at focal sites). Prior use of an investigational monoclonal antibody therapy within 3 months, or prior use of nitrosoureas or mitomycin C within 6 weeks. Patients must have recovered from acute toxicity due to radiotherapy.
* With the exception of alopecia, any unresolved toxicities from prior anti-tumor treatments (excluding corticosteroids) should be no greater than CTCAE (Version 4.0) Grade 1 at the time of study entry.
* Major surgery within 4 weeks prior to entry to the study (excluding placement of vascular access), or minor surgery (excluding tumor biopsies) within 14 days of first dose of study treatment
* Participation in another clinical study with an investigational product during the last 21 days.
* History of hypersensitivity to active or inactive excipients of AZD2014 or drugs with a similar chemical structure or class to AZD2014.
* Exposure to potent or moderate inhibitors or inducers of CYP3A4/5, Pgp (MDR1) and BCRP if taken within the stated washout periods before the first dose of study treatment (see Appendix B)
* Exposure to sensitive or narrow therapeutic range substrates of the drug metabolizing enzymes CYP2C8, CYP2C9, CYP2C19, CYP2D6 or the drug transporters Pgp (MDR1), BCRP, OATP1B1, OATP1B3, OCT1 and OCT2 within the appropriate wash-out period (a minimum of 5 x reported elimination half-life) before the first dose of study treatment (see Appendix B)
* Any haemopoietic growth factors (e.g., filgrastim [granulocyte colony-stimulating factor; G-CSF], sargramostim [granulocyte-macrophage colony-stimulating factor; GM-CSF]) within 14 days prior to receiving study treatment..
* Pre-treatment with other mTOR inhibitors may be allowed and should be discussed for each protocol and tumor type separately
* Current refractory nausea and vomiting, malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
* Previous meningioma progression during treatment with other mTORC1/2 inhibitors (but not mTORC1 inhibitors such as everolimus or other rapalogues)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, severe hepatic impairment, interstitial lung disease (bilateral, diffuse, parenchymal lung disease), uncontrolled chronic renal diseases (glomerulonephritis, nephrotic syndrome, Fanconi Syndrome or renal tubular acidosis), current unstable or uncompensated respiratory or cardiac conditions, uncontrolled hypertension, active bleeding diatheses, active hepatitis B or C infection, known active human immunodeficiency virus (HIV) infection, or psychiatric illness/social situations that would limit compliance with study requirements. Screening for chronic conditions is not required.
* History of other malignancies, except: Malignancy treated with curative intent and with no known active disease present for ≥5 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician, (2) adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, (3) adequately treated carcinoma in situ without evidence of disease, or (4) Gleason 6 prostate cancer under observation.
* Patients who have experienced any of the following procedures or conditions currently or in the preceding 12 months:

  * coronary artery bypass graft
  * angioplasty
  * vascular stent
  * myocardial infarction
  * angina pectoris
  * congestive heart failure New York Heart Association Grade ≥2 ( ventricular arrhythmias requiring continuous therapy)
  * supraventricular arrhythmias including atrial fibrillation, which are uncontrolled
  * haemorrhagic or thrombotic stroke, including transient ischaemic attacks or any other central nervous system bleeding
  * History of drug abuse or alcohol abuse, as judged by the Investigator
* Abnormal echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) at baseline (left ventricular ejection fraction [LVEF] <55%. Appropriate correction to be used if a MUGA is performed.
* Pre-existing renal disease including glomerulonephritis, nephritic syndrome, Fanconi Syndrome or renal tubular acidosis
* Mean resting corrected QT interval (QTc), calculated using Fridericia's formula, > 470 msec obtained from 3 electrocardiograms (ECGs), family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation or Torsade de Pointes within 12 months of the patient entering in the study
* Patients with Diabetes Type I or uncontrolled Type II (HbA1c >8% assessed locally) as judged by the Investigator or Abnormal fasting glucose value defined as >126 mg/dL (>7 mmol/L).
* Concomitant medications known to prolong QT interval, or with factors that increase the risk of QTc prolongation or risk of arrhythmic events (such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age).
* Vaccinated with live, attenuated vaccines within 4 weeks of the first dose of study drug.
* Judgment by the Investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements. Note: patients who are likely to require surgery or radiation for NF2-related tumors during the first year of treatment in the investigator's opinion should not be enrolled on this clinical trial.
* Pregnant women are excluded from this study because AZD2014 is an mTORC1/2 inhibiting agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD2014, breastfeeding should be discontinued if the mother is treated with AZD2014.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD2014. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca, CRO staff, and/or staff at the CPU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Plotkin, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AZD2014
Started | 18
Completed | 6
Not Completed | 12
Not completed — Lack of Efficacy | 3
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | AZD2014
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 41 [18 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Response Rate for Target Meningioma
Description: Number of Target Meningiomas with a Decrease in Tumor Volume of at least 20% Compared with Baseline
Time Frame: up to 24 months
Measure: Count of Units; unit: target meningiomas
Units Other Than Participants: target meningiomas
Arm/Group | AZD2014
Number analyzed (Participants) | 18
Number analyzed (target meningiomas) | 18
target meningiomas | 1

2. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Kaplan-Meier methodology will be used to estimate progression-free survival, with the 95% confidence intervals based on Greenwood's formula.
Time Frame: From date of registration until the date of first documented progression assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AZD2014
Number analyzed (Participants) | 18
months | NA [24 to NA] — The median PFS is "not reached" with a 95% confidence interval of (24 months, infinity)

3. Secondary Outcome: Progression Free Survival at 6 Month
Description: Number of target meningiomas without progression at 6 months. Progression is defined using Response Evaluation In Neurofibromatosis and Schwannomatosis (REiNS) criteria, as a 20% increase in the volume of target meningioma compared with baseline
Time Frame: 6 months of treatment
Measure: Count of Units; unit: target meningiomas
Units Other Than Participants: target meningiomas
Arm/Group | AZD2014
Number analyzed (Participants) | 18
Number analyzed (target meningiomas) | 18
target meningiomas | 16

4. Secondary Outcome: Radiographic Response Rate for Non-target Meningiomas
Description: The response rate is the number of non-target meningiomas with at least 20% decrease in volume compared to the baseline volume.
Time Frame: up to 24 months
Measure: Count of Units; unit: non-target meningiomas
Units Other Than Participants: non-target meningiomas
Arm/Group | AZD2014
Number analyzed (Participants) | 18
Number analyzed (non-target meningiomas) | 14
non-target meningiomas | 2

5. Secondary Outcome: Number of Participants With Grade 3 Adverse Events
Description: Grade 3 adverse events as assessed by CTCAE version 5 guidelines
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | AZD2014
Number analyzed (Participants) | 18
Participants
  Abdominal pain | 1
  Anorexia | 1
  Aspartate aminotransferase increased | 1
  Hypophosphatemia | 10
  Pruritis | 1
  Rash, acneifrom | 1
  Urticaria | 1
  Weight loss | 1

6. Secondary Outcome: Radiographic Response Rate of Vestibular Schwannomas
Description: Radiographic response rate is defined as the proportion of vestibular schwannomas with at least 20% decrease in tumor volume compared to baseline
Time Frame: up to 24 months
Measure: Count of Units; unit: vestibular schwannomas
Units Other Than Participants: vestibular schwannomas
Arm/Group | AZD2014
Number analyzed (Participants) | 18
Number analyzed (vestibular schwannomas) | 16
vestibular schwannomas | 3

7. Secondary Outcome: Disease-Specific Quality of Life
Description: Neurofibromatosis 2 Impact on Quality of Life (NFTI-QOL) questionnaire. The total NFTI-QOL score ranges from 0 to 24. The total NFTI-QOL score is higher in people with higher morbidity.
Time Frame: Baseline, after 3 months of treatment, and off study (up to 24 months)
Population: Analysis population is the participants who completed NFTI-QOL questionnaire at baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | AZD2014
Number analyzed (Participants) | 14
score on a scale
  Baseline | 9 [3 to 17]
  After 3 months: number analyzed (Participants) | 11
  After 3 months | 6 [2 to 16]
  Off study | 8.5 [2 to 20]

8. Secondary Outcome: Vestibular Schwannoma-Specific Quality of Life
Description: Penn Acoustic Neuroma-Quality of Life (PAN-QOL) questionnaire. Scores are normalized to range from 0 to 100 with higher scores indicating better quality of life.
Time Frame: Baseline, after 3 months of treatment, and off study (up to 24 months)
Population: Analysis population includes all participants who completed Pan-QOL questionnaires at baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | AZD2014
Number analyzed (Participants) | 15
score on a scale
  Baseline | 58.9 [38.7 to 81.6]
  After 3 months: number analyzed (Participants) | 12
  After 3 months | 65.3 [28.9 to 84.8]
  Off study: number analyzed (Participants) | 12
  Off study | 56.1 [20.5 to 82.1]

9. Secondary Outcome: Number of Participants With Grade 2 Adverse Events
Description: Grade 2 adverse events as assessed by CTCAE version 5 guidelines
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | AZD2014
Number analyzed (Participants) | 18
Participants
  Abdominal pain | 1
  Anorexia | 2
  Aspartate aminotransferase increased | 2
  Hypophosphatemia | 2
  acute kidney injury | 1
  anemia | 1
  Tachycardia | 1
  Weight loss | 2
  Increased cholesterol | 2
  Creatine phosphokinase increased | 1
  Diarrhea | 6
  dyspareunia | 1
  Fatigue | 2
  Increased triglycerides | 1
  Mucositis | 2
  Nausea | 5
  Vomiting | 1

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | AZD2014
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 7/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2014 (N=18)
Heat stroke (General disorders) | 1
Weight loss (Investigations) | 1
Seizure (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 1
Psychosis (Psychiatric disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2014 (N=18)
Abdominal pain (Gastrointestinal disorders) | 10
Acute kidney injury (Renal and urinary disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
anemia (Blood and lymphatic system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 7
aspartate aminotransferase increased (Investigations) | 5
tachycardia (Cardiac disorders) | 1
dyspepsia (Gastrointestinal disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3
Constipation (Gastrointestinal disorders) | 4
Creatine phosphokinase increased (Investigations) | 1
Diarrhea (Gastrointestinal disorders) | 15
Jaw weakness (Nervous system disorders) | 1
Dry mouth (Gastrointestinal disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 6
Dyspareunia (Reproductive system and breast disorders) | 1
fatigue (General disorders) | 12
Headache (Nervous system disorders) | 2
Hematochezia (Gastrointestinal disorders) | 1
High cholesterol (Metabolism and nutrition disorders) | 3
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hyphophosphatemia (Investigations) | 13
infection (Infections and infestations) | 3
malaise (General disorders) | 1
Difficulty chewing (Nervous system disorders) | 1
mucositis (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 16
Pruritis (Skin and subcutaneous tissue disorders) | 3
Rash, acneiform (Skin and subcutaneous tissue disorders) | 3
amenorrhea (Reproductive system and breast disorders) | 1
Seizure (Nervous system disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
vaginal pain (Reproductive system and breast disorders) | 1
vomiting (Gastrointestinal disorders) | 6
Weight loss (Investigations) | 9
white blood cells decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT02831257/Prot_SAP_000.pdf